CLINICAL TRIAL: NCT02861118
Title: Impact of Co-morbidities on Treatment Response in Inflammatory Bowel Disease: VERNE Study
Brief Title: A Retrospective Observational Study to Assess the Impact of Co-morbidities on Treatment Response in Inflammatory Bowel Disease
Status: Completed | Type: Observational
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Other Study IDs: Vedolizumab-5016
Record Dates: First submitted 2016-08-05; First posted 2016-08-10 (Estimated); Results first posted 2019-08-14 (Actual); Last update posted 2019-08-14 (Actual); Status verified 2019-07

CONDITIONS: Inflammatory Bowel Disease
Keywords: Drug Therapy
MeSH Terms: conditions — Inflammatory Bowel Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Cohort 1: Crohn's Disease: Participants with Crohn's disease who received biological treatment between June 2011 and June 2013.
  Interventions: Other: No Intervention
- Cohort 2: Ulcerative Colitis: Participants with ulcerative colitis who received biological treatment between June 2011 and June 2013.
  Interventions: Other: No Intervention

INTERVENTIONS:
Other: No Intervention

SUMMARY:
The purpose of this study was to evaluate the impact of the co-morbidities profile on treatment response to biological therapy in inflammatory bowel disease (IBD) participants.

DETAILED DESCRIPTION:
This was a retrospective, non-interventional, observational study that included participants diagnosed with ulcerative colitis (UC) or Crohn's disease (CD) who started treatment with biologics between June 2011 and June 2013. The study looked at the impact of the co-morbidities on the treatment response in IBD participants.

The study enrolled 310 patients included both UC and CD patients.

This multicenter trial was conducted in Spain. Investigator collected retrospective data in a single visit from participants who started biologic treatment between June 2011 and June 2013. Time since participants started biological treatment until study visit or until lack of treatment response or until treatment change constituted the reference period for the study.

ELIGIBILITY:
Inclusion Criteria:

* Adult participants (aged ≥18).
* Were diagnosed with UC or CD according to the "World Gastroenterology Organization Practice Guidelines for the Diagnosis and Management of inflammatory bowel disease (IBD) in 2010".
* Who were naive to biologics that started treatment with biologics between June 2011 and June 2013.
* Participants in whom biological treatment was prescribed according to clinical practice.
* Who gave written informed consent.

Exclusion Criteria:

* Were participating in a clinical trial during the study reference period.
* Participant that, according to investigator's criteria was not capable to understand and fill in the study questionnaires or to give written informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Ulcerative colitis (UC) and Crohn's disease (CD) participants who started treatment with biologics between June 2011 and June 2013 will participate in the study.
Sampling Method: Non-Probability Sample
Enrollment: 310 (Actual)
Dates: Start 2016-10-26 (Actual); Primary Completion 2018-04-04 (Actual); Study Completion 2018-04-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (23):
- Spain (23):
  - Santiago de Compostela, A Coruna
  - Huesca, Aragon
  - Alcázar de San Juan, Ciudad Real
  - Girona, Gerona
  - Las Palmas, Gran Canaria
  - Alcorcón, Madrid
  - Fuenlabrada, Madrid
  - Parla, Madrid
  - Pamplona, Navarre
  - Vigo, Pontevedra
  - Gijón, Principality of Asturias
  - Castellon, Valencia
  - Sagunto, Valencia
  - Barakaldo, Vizcaya
  - Barcelona
  - Burgos
  - Ciudad Real
  - Madrid
  - Murcia
  - Santander
  - Seville
  - Valencia
  - Valladolid

IPD SHARING:
Plan to Share IPD: Yes
Takeda makes patient-level, de-identified data sets and associated documents available after applicable marketing approvals and commercial availability have been received, an opportunity for the primary publication of the research has been allowed, and other criteria have been met as set forth in Takeda's Data Sharing Policy (see www.TakedaClinicalTrials.com/approach for details). To obtain access, researchers must submit a legitimate academic research proposal for adjudication by an independent review panel, who will review the scientific merit of the research and the requestor's qualifications and conflict of interest that can result in potential bias. Once approved, qualified researchers who sign a data sharing agreement are provided access to these data in a secure research environment.

REFERENCES:
- [Derived] Marin-Jimenez I, Bastida G, Fores A, Garcia-Planella E, Arguelles-Arias F, Sarasa P, Tagarro I, Fernandez-Nistal A, Montoto C, Aguas M, Santos-Fernandez J, Bosca-Watts MM, Ferreiro R, Merino O, Aldeguer X, Cortes X, Sicilia B, Mesonero F, Barreiro-de Acosta M. Impact of comorbidities on anti-TNFalpha response and relapse in patients with inflammatory bowel disease: the VERNE study. BMJ Open Gastroenterol. 2020 Mar 26;7(1):e000351. doi: 10.1136/bmjgast-2019-000351. eCollection 2020. PMID 32337054

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at the 25 investigative sites in Spain from 26 October 2016 to 04 April 2018.
Pre-assignment Details: Participants with a diagnosis of ulcerative colitis (UC) or Crohn's disease (CD) who started treatment with biologics between June 2011 and June 2013, participated in the study. Total 357 participants were registered, out of which only 310 participants were analyzed.
Period: Overall Study
Arm/Group | Cohort 1: Crohn's Disease | Cohort 2: Ulcerative Colitis
Started | 194 | 116
Completed | 194 | 116
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Analyzed participants included all participants who didn't had screen failure, met all the inclusion criteria and had enough information about response to the biological treatment.
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1: Crohn's Disease | Cohort 2: Ulcerative Colitis | Total
Number analyzed (Participants) | 194 | 116 | 310
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.8 (12.8) | 46.8 (13.3) | 44.9 (13.00)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Male | 103 | 63 | 166
  Female | 90 | 47 | 137
  Not Available | 1 | 6 | 7
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 189 | 108 | 297
  Latin | 3 | 1 | 4
  Gipsy | 1 | 0 | 1
  Arab | 0 | 1 | 1
  Not Available | 1 | 6 | 7
Region of Enrollment [Count of Participants; unit: Participants]
  Spain | 194 | 116 | 310
Working Status [Count of Participants; unit: Participants]
  Employed by Other | 115 | 51 | 166
  Self Employed | 15 | 17 | 32
  Retired | 16 | 16 | 32
  Housework | 12 | 11 | 23
  Unemployed | 17 | 4 | 21
  Student | 6 | 6 | 12
  Permanently Unable to Work | 6 | 3 | 9
  Temporarily Unable to Work | 4 | 1 | 5
  Other | 1 | 1 | 2
  Not Available | 2 | 6 | 8
Level of Education [Count of Participants; unit: Participants]
  Secondary Education | 101 | 46 | 147
  Primary Education | 45 | 30 | 75
  University Education | 42 | 32 | 74
  Uneducated | 4 | 2 | 6
  Not Available | 2 | 6 | 8
Smoking Habits [Count of Participants; unit: Participants]
  Non-smoker | 86 | 70 | 156
  Ex-smoker | 52 | 37 | 89
  Smoker | 55 | 7 | 62
  Not Available | 1 | 2 | 3
Alcohol Abuse [Count of Participants; unit: Participants] — Population: Number analyzed is the number of participants with evaluable data at this baseline measure.
  Participants
    Yes | 4 | 0 | 4
    No | 189 | 114 | 303
    Not Available | 1 | 2 | 3

OUTCOME MEASURES:

1. Primary Outcome: Impact of the Comorbidities Profile in Inflammatory Bowel Disease (IBD) Participants on Lack of Treatment Response to Biological Therapy
Description: Correlation between co-morbidities profile and lack of response, adjusted for sociodemographic and clinical profile of participants, logistic regression models were conducted. Lack of response was reduction of 2 points from baseline in Harvey-Bradshaw Indices (HBI) score for CD or Partial Mayo score (PMS) for UC after 10 weeks treatment with anti-tumour necrosis factor (TNF). HBI included general well-being (0=very well to 4=terrible), abdominal pain (0=none to 3=severe), number of liquid stools/day, abdominal mass (0=none to 3=tender), and complications (8 items; 1 score/item). The total score was sum of sub scores, where score <5=remission, 5-7=mild disease, 8-16=moderate disease and >16-severe disease. PMS included 3 sub-scores: stool frequency (0=normal to 3=>4 stools/day more than normal), rectal bleeding (0=none to 3=passing blood alone), and physician's global assessment (0=Normal to 3=severe). The total score was sum of sub scale scores from 0=normal to 9=severe disease.
Time Frame: Up to 10 weeks after start of treatment with biologics
Population: as for baseline characteristics
Measure: Number (95% Confidence Interval); unit: odds ratio
Groups:
- Participants With Inflammatory Bowel Disease (IBD): Participants with IBD (Crohn's disease and ulcerative colitis) who received biological treatment between June 2011 and June 2013.
Arm/Group | Participants With Inflammatory Bowel Disease (IBD)
Number analyzed (Participants) | 310
odds ratio
  IBD | 0.59 [0.37 to 0.93]
  Corticosteroids | 2.16 [1.25 to 3.73]
  Chronic Obstructive Pulmonary Disease | 2.67 [1.33 to 5.35]
Statistical Analysis 1: Comparison: Participants With Inflammatory Bowel Disease (IBD); IBD; Test type: Other; p = 0.024, Regression, Logistic
Statistical Analysis 2: Comparison: Participants With Inflammatory Bowel Disease (IBD); Corticosteroids; Test type: Other; p = 0.006, Regression, Logistic
Statistical Analysis 3: Comparison: Participants With Inflammatory Bowel Disease (IBD); Chronic Obstructive Pulmonary Disease; Test type: Other; p = 0.006, Regression, Logistic

2. Primary Outcome: Impact of the Comorbidities Profile in IBD Participants on Loss of Treatment Response to Biological Therapy
Description: Correlation between co-morbidities profile and loss of response, adjusted for sociodemographic and clinical profile of participants, logistic regression models were conducted. Loss of response was deﬁned as loss of drug effect along follow up with initial response i.e. reduction of 2 points from baseline in HBI score for CD or PMS for UC after 6 months of treatment with anti-TNF. HBI included general well-being (0=very well to 4=terrible), abdominal pain (0=none to 3=severe), number of liquid stools/day, abdominal mass (0=none to 3=tender), and complications (8 items; 1 score/item). The total score was sum of sub scores, <5=remission, 5-7=mild disease, 8-16=moderate disease and >16=severe disease. PMS score included 3 sub-scores: stool frequency (0=normal to 3=>4 stools/day more than normal), rectal bleeding (0=none to 3=passing blood alone), and physician's global assessment (0=Normal to 3=severe). The total score was sum of sub scale scores ranging from 0=normal to 9=severe disease.
Time Frame: Up to 6 months after start of treatment with biologics
Population: as for baseline characteristics
Measure: Number (95% Confidence Interval); unit: odds ratio
Arm/Group | Participants With Inflammatory Bowel Disease (IBD)
Number analyzed (Participants) | 310
odds ratio
  IBD | 0.58 [0.34 to 0.99]
  Corticosteroids | 2.45 [1.35 to 4.44]
  Myocardial Infarction | 3.30 [1.48 to 7.35]
Statistical Analysis 1: Comparison: Participants With Inflammatory Bowel Disease (IBD); IBD; Test type: Other; p = 0.044, Regression, Logistic
Statistical Analysis 2: Comparison: Participants With Inflammatory Bowel Disease (IBD); Corticosteroids; Test type: Other; p = 0.003, Regression, Logistic
Statistical Analysis 3: Comparison: Participants With Inflammatory Bowel Disease (IBD); Myocardial Infarction; Test type: Other; p = 0.003, Regression, Logistic

3. Secondary Outcome: Impact of the Extraintestinal Manifestations Profile in IBD Participants on Lack of Treatment Response to Biological Therapy
Description: Correlation between extraintestinal manifestations profile and lack of response, adjusted for sociodemographic and clinical profile of participants, logistic regression models were conducted. Lack of response was reduction of at least 2 points from baseline in HBI score for CD or PMS for UC after 10 weeks treatment with TNF. HBI included general well-being (0=very well to 4=terrible), abdominal pain (0=none to 3=severe), number of liquid stools/day, abdominal mass (0=none to 3=tender), and complications (8 items; 1 score/item). The total score was sum of sub scores, where score <5=remission, 5-7=mild disease, 8-16=moderate disease and >16-severe disease. PMS included 3 sub-scores: stool frequency (0=normal to 3=>4 stools/day more than normal), rectal bleeding (0=none to 3=passing blood alone), and physician's global assessment (0=Normal to 3=severe). The total score was sum of sub scale scores from 0=normal to 9=severe disease.
Time Frame: Up to 10 weeks after start of treatment with biologics
Population: as for baseline characteristics
Measure: Number (95% Confidence Interval); unit: odds ratio
Arm/Group | Participants With Inflammatory Bowel Disease (IBD)
Number analyzed (Participants) | 310
odds ratio | 2.08 [1.22 to 3.54]
Statistical Analysis 1: Comparison: Participants With Inflammatory Bowel Disease (IBD); Corticosteroids; Test type: Other; p = 0.007, Regression, Logistic

4. Secondary Outcome: Impact of the Extraintestinal Manifestations Profile in IBD Participants on Loss of Treatment Response to Biological Therapy
Description: Correlation between extraintestinal manifestations profile and loss of response, adjusted for sociodemographic and clinical profile, logistic regression models were conducted. Loss of response was deﬁned as loss of drug effect along follow up with initial response i.e. reduction of 2 points from baseline in HBI score for CD or PMS for UC after 6 months of treatment with anti-TNF. HBI included general well-being (0=very well to 4=terrible), abdominal pain (0=none to 3=severe), number of liquid stools/day, abdominal mass (0=none to 3=tender), and complications (8 items; 1 score/item). The total score was sum of sub scores, <5=remission, 5-7=mild disease, 8-16=moderate disease and >16=severe disease. PMS score included 3 sub-scores: stool frequency (0=normal to 3=>4 stools/day more than normal), rectal bleeding (0=none to 3=passing blood alone), and physician's global assessment (0=Normal to 3=severe). The total score was sum of sub scale scores ranging from 0=normal to 9=severe disease.
Time Frame: Up to 6 months after start of treatment with biologics
Population: as for baseline characteristics
Measure: Number (95% Confidence Interval); unit: odds ratio
Arm/Group | Participants With Inflammatory Bowel Disease (IBD)
Number analyzed (Participants) | 310
odds ratio
  Corticosteroids | 2.57 [1.43 to 4.61]
  Skin Disease | 2.73 [1.42 to 5.25]
Statistical Analysis 1: Comparison: Participants With Inflammatory Bowel Disease (IBD); Corticosteroids; Test type: Other; p = 0.002, Regression, Logistic
Statistical Analysis 2: Comparison: Participants With Inflammatory Bowel Disease (IBD); Skin Disease; Test type: Other; p = 0.003, Regression, Logistic

5. Secondary Outcome: Percentage of IBD Participants With Comorbidities
Description: Participants with CD and UC along with comorbidities were reported. Comorbidity referred to the presence of co-existing or additional diseases with reference to an initial diagnosis or with reference to the index condition.
Time Frame: Day 1
Population: Analyzed participants included all participants who didn't had screen failure, met all the inclusion criteria and had enough information about response to the biological treatment. Number analyzed is the number of participants with evaluable data at the given time-point.
Measure: Number; unit: percentage of participants
Arm/Group | Cohort 1: Crohn's Disease | Cohort 2: Ulcerative Colitis
Number analyzed (Participants) | 194 | 116
percentage of participants
  Myocardial Infarction: number analyzed (Participants) | 185 | 114
  Myocardial Infarction | 2.2 | 0.9
  Congestive Heart Failure: number analyzed (Participants) | 185 | 114
  Congestive Heart Failure | 1.6 | 0.9
  Peripheral Vascular Disease: number analyzed (Participants) | 185 | 114
  Peripheral Vascular Disease | 1.6 | 0.0
  Cardiovascular Disease: number analyzed (Participants) | 185 | 114
  Cardiovascular Disease | 0.5 | 2.6
  Chronic Obstructive Pulmonary Disease: number analyzed (Participants) | 185 | 114
  Chronic Obstructive Pulmonary Disease | 3.2 | 4.4
  Connective Tissue Disease: number analyzed (Participants) | 185 | 114
  Connective Tissue Disease | 2.7 | 3.5
  Peptic Ulcer Disease: number analyzed (Participants) | 185 | 114
  Peptic Ulcer Disease | 0.5 | 0.9
  Mild Chronic Hepatopathy: number analyzed (Participants) | 185 | 114
  Mild Chronic Hepatopathy | 1.1 | 3.5
  Diabetes Mellitus: number analyzed (Participants) | 185 | 114
  Diabetes Mellitus | 0.5 | 5.3
  Diabetes with Lesions in Target Organs: number analyzed (Participants) | 185 | 114
  Diabetes with Lesions in Target Organs | 0.0 | 0.9
  Solid Tumor: number analyzed (Participants) | 185 | 114
  Solid Tumor | 2.2 | 0.9
  Leukemia: number analyzed (Participants) | 185 | 114
  Leukemia | 0.0 | 0.9
  Lymphoma: number analyzed (Participants) | 185 | 114
  Lymphoma | 0.5 | 0.0
  Moderate-Severe Chronic Hepatopathy: number analyzed (Participants) | 185 | 114
  Moderate-Severe Chronic Hepatopathy | 0.5 | 0.0

6. Secondary Outcome: Percentage of CD Participants With Comorbidities According to the Level of IBD Severity
Description: Participants with CD were classified into IBD severe or non-severe at baseline based on the HBI scores according the following criteria:- HBI includes general well-being (0=very well to 4=terrible), abdominal pain (0=none to 3=severe), number of liquid stools per day, abdominal mass (0=none to 3=tender), and complications (8 items; 1 score/item). The total score is sum of sub scores, score <5=remission, 5-7=mild disease, 8-16=moderate disease and >16=severe disease.
Time Frame: Day 1
Population: as for outcome 5
Measure: Number; unit: percentage of participants
Arm/Group | Cohort 1: Crohn's Disease
Number analyzed (Participants) | 194
percentage of participants
  Non-Severe Disease: number analyzed (Participants) | 162
  Non-Severe Disease | 62.4
  Severe Disease: number analyzed (Participants) | 162
  Severe Disease | 8.3

7. Secondary Outcome: Percentage of UC Participants With Comorbidities According to the Level of IBD Severity
Description: Participants with UC were classified into IBD severe or non-severe at baseline based on the PMS scores according the following criteria:- PMS score includes 3 sub-scores: stool frequency (0=normal to 3=>4 stools/day more than normal), rectal bleeding (0=none to 3=passing blood alone), and physician's global assessment (0=Normal to 3=severe). The total score is sum of sub scale scores ranging from 0=normal to 9=severe disease.
Time Frame: Day 1
Population: as for outcome 5
Measure: Number; unit: percentage of participants
Arm/Group | Cohort 2: Ulcerative Colitis
Number analyzed (Participants) | 116
percentage of participants
  Non-Severe Disease: number analyzed (Participants) | 108
  Non-Severe Disease | 37.6
  Severe Disease: number analyzed (Participants) | 108
  Severe Disease | 91.7

ADVERSE EVENTS:
Time Frame: Time since participants started biological treatment until study visit (Day 1)
Description: At each visit the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment.
Arm/Group | Cohort 1: Crohn's Disease | Cohort 2: Ulcerative Colitis
All-Cause Mortality (participants affected / at risk) | 0/194 | 0/116
Serious Adverse Events (participants affected / at risk) | 0/194 | 1/116
Other Adverse Events (participants affected / at risk) | 0/194 | 0/116
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1: Crohn's Disease (N=194) | Cohort 2: Ulcerative Colitis (N=116)
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The first study related publication will be a multi-center publication submitted within 24 months after conclusion or termination of a study at all sites. After such multi site publication, all proposed site publications and presentations will be submitted to sponsor for review 60 days in advance of publication. Site will remove Sponsor confidential information unrelated to study results. Sponsor can delay a proposed publication for another 60 days to preserve intellectual property.

DOCUMENTS (2):
  • Statistical Analysis Plan (2017-02-15): https://cdn.clinicaltrials.gov/large-docs/18/NCT02861118/SAP_000.pdf
  • Study Protocol (2016-04-13): https://cdn.clinicaltrials.gov/large-docs/18/NCT02861118/Prot_001.pdf